CLINICAL TRIAL: NCT01099384
Title: Tobacco Cessation Treatment for Alaska Native Youth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Yukon Kuskokwim Health Corporation (Other)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-003981; R01DA025156 (NIH)
Record Dates: First submitted 2010-04-02; First posted 2010-04-07 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral: written self-help materials (Active Comparator): Behavioral: written self-help materials
  Interventions: Behavioral: Written self-help materials
- Group behavioral counseling (Experimental): Group behavioral counseling, weekend program
  Interventions: Behavioral: Group behavioral counseling

INTERVENTIONS:
Behavioral: Written self-help materials — Written materials to help adolescents stop tobacco use
  Other Names: Control condition
  Arms: Behavioral: written self-help materials
Behavioral: Group behavioral counseling — group behavioral counseling (2 day weekend program)
  Other Names: intervention condition
  Arms: Group behavioral counseling

SUMMARY:
Tobacco use among adolescents is a major public health problem in the United States. The prevalence of tobacco use among adolescents is currently highest among American Indians and Alaska Natives. Among Alaska Natives residing in the Yukon-Kuskokwim (Y-K) Delta region of western Alaska, approximately 29% of 11-14 year olds, and 63% of 15-18 year olds, use tobacco. No prior work has evaluated tobacco cessation interventions for Alaska Native adolescents.

This proposal builds on the investigators successful partnership and 7 year track record of collaboration with the Y-K Delta Alaska Native community. The objective of this proposal is to develop and pilot test a novel, culturally-appropriate, behavioral treatment approach for tobacco cessation among Y-K Delta Alaska Native adolescents ages 12 to 17. The behavioral intervention will include an initial, 2 day, group-based program with follow-up support for 6 weeks. Social cognitive (learning) theory is the conceptual basis for the proposed intervention. The investigators expect that as a result of this stage I project, the investigators will have developed a replicable, feasible, and acceptable intervention, the efficacy of which can be tested in future large-scale randomized clinical trials.

This project will take place in two phases. In phase 1, the investigators will develop the intervention with feedback from a teen advisory group, and develop a counselor manual. Follow-up strategies will also be developed, pilot-tested, and refined. Twenty adolescents will complete the protocol, which will be refined in an iterative manner based on feedback from participants and counselors. Phase 2, consisting of a pilot clinical trial, will apply a group-randomized design with assessments at weeks 0 (baseline), 6, and 26. Eight villages will be randomized to receive either the behavioral intervention or control condition (written self-help materials + quitline referral). Ten adolescents will be enrolled from each village, for a total of 80 participants. The investigators will assess the feasibility and acceptability of the intervention, as determined by qualitative ratings of treatment acceptability, and recruitment and retention rates. The investigators will estimate the magnitude of the effect of the intervention compared to the control condition on the biochemically confirmed tobacco abstinence rate at weeks 6 and 26, and estimate the intra-class correlation coefficient (ICC). At week 6, the investigators will evaluate the effect of the intervention on changes from baseline on perceived social support, self-efficacy for stopping tobacco use, and other mechanisms of change consistent with the investigators theoretical framework. The overall health related objective is to develop effective treatment programs for Alaska Native youth that will ultimately reduce their risk of tobacco-related disease.

ELIGIBILITY:
Inclusion Criteria:

1. Alaska Native
2. is from one of the targeted villages
3. is between 12-17 years of age
4. provides written assent
5. provides written parental consent
6. self-reports daily use of Iqmik, commercial ST, and/or cigarette smoking during the past 7 days, with current tobacco use status verified with a NicAlert salivary cotinine test strip value of >0
7. is willing to make a quit attempt
8. is willing and able to participate in all aspects of the study
9. has access to Web/e-mail and a working telephone.

Exclusion Criteria:

1. the adolescent is not able to fully participate in the intervention or would potentially pose harm to self or other group participants, and/or disrupt the group process (e.g., if subject is intoxicated at screening)
2. depression score of >16 as assessed by the Center for Epidemiological Studies Depression Scale (CES-D; Radloff, 1977)
3. current (past 3 months) participation in any tobacco pharmacological or behavioral treatment
4. another adolescent from the same household has enrolled.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | Assessed at the time of screening

SECONDARY OUTCOMES:
Biochemically confirmed tobacco abstinence | Assessed at Week 6 (End of Treatment)
Study retention | Assessed at week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Yukon Kuskokwim Health Corporation, Bethel, Alaska, United States